CLINICAL TRIAL: NCT04880018
Title: Clinical Validation Plan of Capsular Tension Ring
Acronym: CVPOCTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyebright Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB/JS-QD-123; 2015QXNL002 (Other: Zhongshan Ophthalmic Center, Sun Yat-sen University)
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Intraocular Lens Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsular Tension Ring from Eyebright Medical Technology (Beijing) Co., Ltd (Experimental): Specification model: CTR1109、CTR1210、CTR1311、CTR1412、CTR1513 Manufacturer: Eyebright Medical Technology (Beijing) Co., Ltd.
  Interventions: Device: Capsular Tension Ring
- Capsular Tension Ring from Carl Zeiss Medical Technology Co., Ltd (Active Comparator): Specification model: TENSIOBAG 10、TENSIOBAG 11、TENSIOBAG 12、TENSIOBAG 13、TENSIOBAG14 Manufacturer: Carl Zeiss Medical Technology Co., Ltd.
  Interventions: Device: Capsular Tension Ring

INTERVENTIONS:
Device: Capsular Tension Ring — Experimental group uses Capsular Tension Ring from Eyebright Medical Technology (Beijing) Co., Ltd;control group uses Capsular Tension Ring from Carl Zeiss Medical Technology Co., Ltd

SUMMARY:
Through follow-up for 1 year or more, the safety and effectiveness of the Capsular Tension Ring produced by Eyebright Medical Technology (Beijing) Co., Ltd. were verified, which is used for intraocular lens implantation in aphakic eyes after lens extraction to maintain capsular integrity, prevent posterior capsular wrinkle and resist capsular shrinkage.

The clinical validation plan will be implemented after being approved by the Ethics Committee; the trial data of all cases before the 6-month visit period will be counted, and the statistical report, summary report and sub-center summary will be issued. The summary report and sub-center summary will be submitted to the CFDA for product registration.

DETAILED DESCRIPTION:
According to the principle of "Quality management standard for clinical trials of medical devices" issued by CFDA, a multi-center, randomized, open, positive product, parallel controlled trial design was adopted to evaluate the safety and effectiveness of the Capsular Tension Ring produced by Eyebright Medical Technology (Beijing) Co., Ltd.

Considering the progress of clinical verification and the reliability of the conclusion, the multi-center trial design was adopted in this clinical verification. Multi-center clinical trials can collect more cases in a short time, and cover a wide population of cases, which avoids the limitations of a single research, and the conclusions can have a wider significance and greater credibility. In order to demonstrate the effectiveness and safety of the product, and to verify whether the product has the same efficacy and safety as the marketed product, a positive product and a parallel controlled trial design were selected for the validation; The "Capsular Tension Ring" produced by Carl Zeiss, with the same material, structure, design, implantation mode and location, and indications, was selected as the positive parallel control product, and the clinical trial was conducted simultaneously with the validation product. In view of the fact that this clinical trial is a comparative research of positive products and parallel controls, in order to ensure the comparability of cases in each group, avoid bias caused by various factors in the design, execution, and analysis of the clinical trial. This clinical verification adopts a randomization method and uses a central random system to achieve dynamic randomization to ensure that cases are evenly allocated to the test group or the control group. Due to the variety of product specifications in this clinical verification, the use of the verification product and the reference substance is slightly different. This verification cannot be double-blind, so an open clinical trial design is adopted.

Based on the above considerations and adhering to the scientific principle, in order to verify the safety and effectiveness of the Capsular Tension Ring produced by Eyebright, a multi-center, randomized, open, positive product, parallel controlled trial method was adopted in this clinical verification.

At the same time, 120 cases of cataract patients were selected according to the statistical requirements. After screening and examination, those who met the inclusion criteria were selected for validation. Surgical treatment and implantation of validation or control products were performed. Clinical follow-up evaluation was planned at 1-2 days, 1 week, 1 month, 3 months, 6 months and 1 year after operation. The percentage of patients whose best corrected visual acuity reached 20/40 at 6 months after operation was taken as the main efficacy indicator; At the same time, observe the visual acuity, optometry results, intraocular pressure, lens eccentricity, capsule shrinkage, etc. after 1~2 days, 1 week, 1 month, 3 months, 6 months and 1 year or more after operation; The main safety indicators are the incidence of complications, adverse events and serious adverse events during the observation period, and adverse events and serious adverse events related to the validated device.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old, no gender limit;
2. For cataract patients who are expected to undergo phacoemulsification + Capsular Tension Ring and intraocular lens implantation, the hardness of the surgical eye nucleus is 1 to 3;
3. Be able to understand the purpose of the trial, voluntarily participate in and sign informed consent form by the patient himself or his legal guardian.

Exclusion Criteria:

Inclusion criteria

1. Over 18 years old, no gender limit;
2. For cataract patients who are expected to undergo phacoemulsification + Capsular Tension Ring and intraocular lens implantation, the hardness of the surgical eye nucleus is 1 to 3;
3. Be able to understand the purpose of the trial, voluntarily participate in and sign informed consent form by the patient himself or his legal guardian.

Exclusion criteria

1. The surgical eye has other ocular diseases, those with Capsular Tension Ring implantation or intraocular operation contraindications, such as binocular congenital cataracts, microphthalmia, children under the age of 12 months, corneal dystrophy or endothelial cell insufficiency, chronic uveitis, active ocular diseases (Diabetic retinopathy active stage, uncontrollable glaucoma), fragile capsular bag, zonular rupture exceeding 120 degrees, etc.
2. Accompanied by severe or unstable heart, liver, kidney, lung, endocrine (including thyroid insufficiency), blood, mental and nerve dysfunction and other diseases;
3. The surgical eye has had retinal detachment or retinopathy;
4. Patients with congenital cataracts undergoing operation;
5. Those whose electrocardiogram examination or laboratory examination results suggest surgical contraindications;
6. Those who are unsupervised or cannot follow the doctor's advice;
7. Those with a history of intraocular operation in the last 3 months;
8. It is estimated that the best corrected distance visual acuity after operation is less than 20/40;
9. Those who need combined eye operation;
10. Participated in clinical trials of other drugs or medical devices within 30 days before screening;
11. Patients who are using or need to use ocular or systemic drugs during the research period that may affect their visual acuity;
12. Pregnant or breastfeeding women;
13. Those who have been judged by the researcher to ignore the function of the contralateral eye;
14. The researcher judges that the patient is not suitable for other situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Best corrected distance visual acuity | At 6 months after operation
  The percentage of eyes whose best corrected distance visual acuity reached 20/40 at 6 months after operation

SECONDARY OUTCOMES:
Best corrected distance visual acuity, uncorrected distance visual acuity | In 1~2 days, 1 week, 1 month, 3 months, 6 months, 1 year
  Visual acuity in 1~2 days, 1 week, 1 month, 3 months, 6 months, 1 year
Diopter | In 1~ 2 days, 1 week, 1 month, 3 months, 6 months, 1 year
  Dioptric power of 1 to 2 days, 1 week, 1 month, 3 months, 6 months, 1 year
The intraocular lens eccentricity | In 1~ 2 days, 1 week, 1 month, 3 months, 6 months, 1 year
  Eccentricity of intraocular lens of 1 to 2 days, 1 week, 1 month, 3 months, 6 months, 1 year
The capsular shrinkage | In 1~ 2 days, 1 week, 1 month, 3 months, 6 months, 1 year
  Capsule contraction of 1 to 2 days, 1 week, 1 month, 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ye, PhD, Study Director; Yong Zhong, PhD, Study Director; Qi Han, PhD, Study Director — Tianjin Medical University General Hospital; Jun Fang, PhD, Study Director — Daqing oilfield general hospital; Ayong Yv, PhD, Study Director — Opto-optic Hospital of Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No